CLINICAL TRIAL: NCT06883435
Title: A Prospective Comparative Study Between Percutaneous Cannulated Screws and Open Reduction and Internal Fixation in Treatment of Displaced Isolated Medial Malleolar Fractures
Brief Title: Percutaneous Cannulated Screws Versus Open Reduction and Internal Fixation in the Treatment of Displaced Isolated Medial Malleolar Fractures in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khalaf fathy elsayed Ahmed, Principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-23-03-09PD
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Medial Malleolus
Keywords: Isolated medial malleolar fractures, Displaced, Percutaneous fixation, open reduction, Cannulated screws
MeSH Terms: interventions — Open Fracture Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- closed reduction and percutaneous ﬁxation (CRPF) (Experimental): percutaneous cannulated screws fixation of medial malleolus
  Interventions: Procedure: closed reduction and percutaneous ﬁxation of medial malleolus
- open reduction and internal fixation (ORIF) (Experimental): Open reduction and screw fixation of medial malleolus
  Interventions: Procedure: open reduction and screw fixation of medial malleolus

INTERVENTIONS:
Procedure: closed reduction and percutaneous ﬁxation of medial malleolus — No incision is made for fracture reduction, a pointed reduction clamp is applied to reduce the fracture, two 4 mm partially threaded cannulated cancellous screws are inserted over guide wires through stab incisions. Fluoroscopy is used to assess reduction.
  Arms: closed reduction and percutaneous ﬁxation (CRPF)
Procedure: open reduction and screw fixation of medial malleolus — An incision is made over the fracture; the MM fracture is reduced under direct vision. fixation is performed with two 4mm cannulated partially threaded cancellous screws. fluoroscopy is used to confirm reduction.
  Arms: open reduction and internal fixation (ORIF)

SUMMARY:
The aim of this prospective randomized controlled trial is to compare the functional and radiographic outcomes of closed reduction and percutaneous cannulated screws fixation and ORIF in treatment of displaced isolated medial malleolar fractures.

DETAILED DESCRIPTION:
Medial malleolar (MM) fractures occur in about 50% of all ankle fractures, and may occur as isolated MM fractures or as part of a bi- or tri-malleolar ankle fractures.

MM fractures may occur following road traffic accident, twisting injury to ankle, assault, and falling from height.

When MM fractures occurring as a part of a bi- or tri-malleolar ankle fractures, MM fractures are typically treated with surgical fixation. Isolated non-displaced MM fractures can be treated conservatively by below knee cast application. Displaced isolated MM fractures are usually treated surgically.

Many fixation techniques for MM fractures have been proposed including; unicortical partially threaded compression screws, bicortical fully threaded screws, buttress or neutralization plates, and tension band wiring. The choice of a particular fixation technique depends on the fracture geometry and the extent of comminution. Surgical procedures can be done by open reduction internal fixation (ORIF) or closed reduction percutaneous fixation.

In comparison to an ORIF, a percutaneous approach to MM fractures have potential advantages of decreased surgical morbidity, decreased postoperative pain, and decreased risk of wound complications. However, without direct fracture site visualization, it is possible that acceptable reduction could be hindered, leading to higher rates of nonunion and malunion. Some studies have shown that even in unstable medial malleolus fractures percutaneous screw fixation is excellent technique.

There is dilemma in the existing literature which treatment method is better for MM fractures management. Up to my knowledge, there is no comparative prospective study of ORIF versus percutaneous approach in surgical treatment of isolated medial malleolar fractures.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with closed, displaced (˃2mm), isolated medial malleolar fractures of Herscovici type B or C.

Exclusion Criteria:

* comminuted fractures, open fractures, bi-, tri-, or quadri-malleolar ankle fractures, associated syndesmotic or lateral collateral ligament injuries, skeletally immature patients, any other ipsilateral lower limb fractures, or previously fractured ankle.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
AOFAS (American association of foot and ankle society) ankle-hind foot score | Baseline
  American association foot and ankle society score for foot and ankle conditions

SECONDARY OUTCOMES:
Foot and ankle ability measure (FAAM) | baseline
  Patient reported outcome measure for foot and ankle condition
visual analogue scale (VAS) | baseline
  method of pain assessment

CONTACTS AND LOCATIONS:
Locations (1):
- SohagU, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed KFE. Percutaneous versus open cannulated screws fixation for displaced isolated medial malleolar fractures in adults: a randomized controlled clinical trial. Arch Orthop Trauma Surg. 2025 Jul 25;145(1):385. doi: 10.1007/s00402-025-06000-w. PMID 40711571